CLINICAL TRIAL: NCT00177684
Title: Pharmacokinetic Profiles of Inhaled Lipid Complex Amphotericin B (Abelcet ®)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Enzon Pharmaceuticals, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB # 0407015
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2008-12-17 (Estimated); Status verified 2008-12

CONDITIONS: Lung Transplantation; Fungal Infections
MeSH Terms: conditions — Mycoses | interventions — Amphotericin B

INTERVENTIONS:
Drug: Amphotericin B

SUMMARY:
The purpose of this study is to determine the optimal delivery system for the nebulization of the lipid complex amphotericin B (Abelcet ®) in lung transplant recipients who are positive for invasive aspergillosis (IA) in their lungs. Additionally, the investigators hope to determine the concentrations of amphotericin B achieved in the epithelial lining fluid, and serum with the administration of four days of lipid complex of amphotericin B (Abelcet ®) (QD) via aerosolized nebulization

DETAILED DESCRIPTION:
Subject's visit for teaching and administration of the first dose of aerosolized liposomal Amphotericin will be performed at the specified intervals before the scheduled bronchoscopy.

Subject will receive first dose of the aerosolized liposomal amphotericin under direct supervision of physician and study coordinator. This visit will last approximately 2 hours.

Subject's spirometry will be performed before (standard of care) and after the administration (research related) of first dose aerosolized liposomal amphotericin. Each spirometry measurement takes approximately 1 hour. Prior to administration, blood pressure and heart rate will be obtained.

In the absence of any significant side effect of the aerosolized liposomal amphotericin (e.g., wheezing, shortness of breath, drop in FEV1 > 15%, the remaining three doses will be dispensed to the patient through pharmacy. The subject will be instructed on how to measure his/her peak flow rate before and after taking the aerosolized liposomal amphotericin. (approximately 1 hour) A 24 hr study pager number will be given to subjects to contact the investigators in case of development of side effects such as shortness of breath, wheezing, heaviness in the chest.

The study coordinator will contact the subject daily to ensure the compliance with the aerosolized liposomal amphotericin administration and monitor any untoward effects. This phone contact will not take longer than 10 minutes of the participant's time.

Drug administration: Subjects will be dispensed vials of ABELCET ® and will be taught by the study coordinator/investigators to draw drug from the vial to nebulizer. Detailed written instructions will also be provided to the subjects. In addition subjects will prove the comprehension of the instructions by demonstrating the procedure, to the study coordinator during initial visit. The description for the patient is as follows "Before administering the drug via nebulization, shake the vial gently until there is no evidence of any yellow sediment at the bottom. Withdraw the appropriate dose of ABELCET ® from the required number of vials into one or more sterile syringes using an 18-gauge needle. Remove the needle from each syringe filled with ABELCET ® and replace with the 5-micron filter needle supplied with each vial. Put no more than 7 ml of ABELCET ® in the nebulizer and inhaled over a period of 15 minutes. Continue the inhalation process until whole the amount is used up. Repeat the procedure with additional drug if your doctor has prescribed more drug for you". Aero Eclipse Nebulizer and Devilbliss 8650D compressor will be used for the study.

ELIGIBILITY:
Inclusion Criteria:

* Male and female lung transplant recipients at University of Pittsburgh Medical Center ≥ 18yrs of age will be eligible for the study. Subjects HIV status will not determine the exclusion from study.

Exclusion Criteria:

* Pregnant women or women who are currently breast-feeding an infant
* Hypersensitive to amphotericin deoxycholate or lipid complex amphotericin B (Abelcet ®)
* Have a documented fungal infection
* Receipt of inhalational or IV amphotericin B within last 30 days
* Have a Temp ≥ 38ºC
* Hypoxemic (pulse oximeter < 92% at room air.)
* On mechanical ventilator

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48
Dates: Start 2004-09; Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
To determine the optimal delivery system for the nebulization of the lipid complex amphotericin B (Abelcet ®).

SECONDARY OUTCOMES:
To determine the concentrations of amphotericin B achieved in the epithelial lining fluid, and serum with the administration of a four days of lipid complex of amphotericin B (Abelcet ®) (QD) via aerosolized nebulization in lung transplant recipients.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Ludwig, Study Director — Enzon Pharmaceuticals, Inc.
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Husain S, Capitano B, Corcoran T, Studer SM, Crespo M, Johnson B, Pilewski JM, Shutt K, Pakstis DL, Zhang S, Carey ME, Paterson DL, McCurry KR, Venkataramanan R. Intrapulmonary disposition of amphotericin B after aerosolized delivery of amphotericin B lipid complex (Abelcet; ABLC) in lung transplant recipients. Transplantation. 2010 Dec 15;90(11):1215-9. doi: 10.1097/TP.0b013e3181f995ea. PMID 20881664